CLINICAL TRIAL: NCT03781154
Title: Predictors of Physical Activity Maintenance in Colorectal Cancer Survivors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Cancer Society, Inc. (Other); Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-2436.cc; 131629-MRSG-18-021- 01-CPPB (Other: American Cancer Society)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
Keywords: Physical activity; Survivors; Maintenance; Personal Training; Group Mediated Cognitive Behavior
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will be prospectively assigned or allocated to either the group-based exercise intervention or control group for 12 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI and study staff conducting assessments at study visits will be blinded to study arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based exercise (Experimental): Virtually-delivered supervised exercise sessions will take place twice per week for approximately one hour, and include aerobic, muscular strength and endurance, balance, and flexibility components.
  Interventions: Behavioral: Group Exercise
- Control Group (No Intervention): A physical activity education control group

INTERVENTIONS:
Behavioral: Group Exercise — Patients will exercise in a virtual group for 60 minutes, twice a week. Five social-cognitive theory-based discussion sessions with the group, and group exercise instructor will be held throughout the course of the intervention, lasting 30 to 60 minutes. The goal of these sessions is to enhance long-term physical activity behavior change.
  Arms: Group-based exercise

SUMMARY:
This study is a two-arm trial, comparing the effects of a virtual 12-week group-based exercise intervention vs. control group on physical activity, physical fitness, and quality of life in colorectal cancer survivors, and explore multi-level determinants of physical activity maintenance, 6-months after intervention completion.

DETAILED DESCRIPTION:
Participants will be prospectively assigned or allocated to either a the exercise intervention or a control group for 12-weeks. The control group will be provided with an informational handout from the American Cancer Society describing exercise recommendations and guidelines for cancer survivors. At the end of the study, control group participants will be offered compensation for participation in a community-based cancer specific exercise program (e.g., BfitBwell, Fit Cancer, Livestrong at the YMCA). Supervised exercise sessions will take place twice per week for approximately one hour, and include aerobic, muscular strength and endurance, balance, and flexibility components. Sessions will be delivered synchronously (i.e., in real-time/live) via Zoom. Exercise will be individualized based on the results of baseline fitness assessments and medical history. The intervention will also include virtual, group-based discussion sessions which operationalize behavior change techniques to increase physical activity. Discussion sessions will take place in the same groups, synchronously, via Zoom.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Fluent in English
3. Have access to a computer or phone with internet and a camera
4. Stated willingness to comply with all study procedures and be available for the duration of the study
5. Be a male or female aged 40 years or older at time of diagnosis
6. Histologically confirmed cancer of the colon or rectum (stages II-IV) if treated with curative intent, and no current evidence of metastatic disease
7. Completed resection or other surgery 3-24 months prior to enrollment
8. Received chemotherapy and/or radiation therapy within the previous year, with at least 1 cycle of intended chemotherapy completed (does not need to complete all cycles). No plans for additional chemotherapy or radiation therapy.

Exclusion Criteria:

1. Current evidence of metastatic disease
2. Existing participation in ≥150 minutes per week of at least moderate intensity PA
3. Known contraindications for exercise or not able to safely participate in exercise
4. Pregnant women (no testing required)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Physical Activity | From baseline to 12-weeks, and 6 months post intervention
  Compare the effects of a 12-week physical activity intervention delivered in group versus control group, on physical activity. Physical activity will be measured with a self-report questionnaire (duration and frequency of moderate and vigorous physical activity) and accelerometer.

SECONDARY OUTCOMES:
Physical Fitness: Aerobic | From baseline to 12-weeks and 6-months post intervention
  Aerobic fitness will be assessed with a submaximal, graded exercise test on a motorized, calibrated treadmill. Muscular Strength & Endurance will be assessed by multiple repetition maximum (1RM) plate loaded seated bench press and leg press, and by the number of full stands from a chair, and the number of bicep curls (holding a hand weight of 5lbs) that can be completed in 30 seconds.
Physical Fitness: Strength and Endurance | From baseline to 12-weeks and 6 months post intervention
  Muscular strength & endurance will be assessed by various weight training activities.
Body Composition | From baseline to 12-weeks 6 months post intervention
  Assessed by waist circumference
Body Composition | From baseline to 12 weeks
  Assessed by the combination of lean mass and fat mass via Dual-Energy X-ray Absorptiometry (DEXA)
Sleep Quality | From baseline to 12 weeks
  Assessed by a self-report measure of sleep quality using the Pittsburg Sleep Quality Index (PSQI) and through the Actiwatch, which is a wrist-worn monitor that records movement and light exposure.
Quality of Life Assessment | From baseline to 12 weeks and 6 months post intervention
  Assessed by a quantitative self-report questionnaire (Functional Assessment of Cancer Therapy-Colorectal (FACT-C)

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, MD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - University of Colorado Denver, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Colorado State University, Fort Collins, Colorado
  - Harmony Campus, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bachman SL, Gomes E, Aryal S, Cella D, Clay I, Lyden K, Leach HJ. Do Measures of Real-World Physical Behavior Provide Insights Into the Well-Being and Physical Function of Cancer Survivors? Cross-Sectional Analysis. JMIR Cancer. 2024 Jul 15;10:e53180. doi: 10.2196/53180. PMID 39008350